CLINICAL TRIAL: NCT04464330
Title: Biomechanical Mechanism of the Change of the Gait Touch Information After ACL Rupture
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OR004
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; gait analysis; plantar pressure; multi-body dynamics modeling
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior Cruciate Ligament injury and reconstruction group: According to the previous clinical diagnosis, patients who has suffered the Anterior Cruciate Ligament injury.
  Interventions: Other: no intervention
- normal control group: According to the previous clinical diagnosis, volunteers who has never suffered the lower extremity sports injuries.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study, with no intervention

SUMMARY:
High incidence rate of knee osteoarthritis and gait analysis are important for early assessment of biomechanics. ACL injury is an ideal clinical model for studying knee osteoarthritis.

To clarify the mechanism between the biomechanical status of knee joint and the change of gait touch information, and to provide scientific basis for quantifying and evaluating the biomechanical status of knee joint in dynamic load-bearing state.

DETAILED DESCRIPTION:
The purpose of this study is to identify the characteristics of the disease, diagnose the disease by computer and evaluate the rehabilitation based on gait touch information after ACL rupture and reconstruction, combined with the methods of multi-body dynamics, machine learning and biomechanics analysis. Methods: 55 healthy volunteers, 55 patients with ACL rupture were recruited. Three dimensional gait analysis and dynamic plantar pressure were used to test the kinematic and dynamic data of lower limbs and gait touch information when walking, jogging, stopping and jumping, and running side cutting.

Outcome evaluation indexes and statistical methods:

the following indexes were measured repeatedly by two factor ANOVA method, and the left and right sides and different rehabilitation time were used as the variables of repeated measurement: the biomechanics of the lower limb joint and the change of the biological characteristics of gait touch information were analyzed. To study the biomechanical status of different knee joints and the mechanism of the change of gait touch information. Finally, based on the information of gait touch, a biomechanical evaluation model of knee joint during walking or jogging is established, which provides the exact basis for quantifying and evaluating the biomechanical state of knee joint under the dynamic load-bearing state of gait touch information.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital.
* With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures).
* All participants have no known disorders or diseases other than ACL rupture.

Exclusion Criteria:

* Cognitive impairment
* Other injuries affecting movement performance.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion criteria: Age: 18-35 years old. Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital. With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures). All participants have no known disorders or diseases other than ACL rupture.
  Exclusion criteria: Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
walking speed | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
knee flexion angle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee flexion in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | On the day of enrollment.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100. The higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No